CLINICAL TRIAL: NCT03338192
Title: Racial and Socioeconomic Differences in Chronic Low Back Pain
Brief Title: Examining Racial and SocioEconomic Disparities (ERASED) in Chronic Low Back Pain Study
Acronym: ERASED
Status: Completed | Type: Observational
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Principal Investigator, Burel Goodin, Principal Investigator, University of Alabama at Birmingham
Other Study IDs: F170119003; R01MD010441 (NIH)
Record Dates: First submitted 2017-11-07; First posted 2017-11-09 (Actual); Results first posted 2025-03-30 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Back Pain Lower Back Chronic
Keywords: Low back pain; Chronic pain; Health disparities in chronic low back pain
MeSH Terms: conditions — Low Back Pain; Chronic Pain

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Specimens will be labeled with unique identifiers (subject numbers) that correspond to each separate participant. Blood samples will be processed for serum and plasma and stored at -80 and then used to detect levels of Vitamin D, C-reactive protein and Oxytocin.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- African American/Black QST: This group will consist of a full range of socioeconomic status in African American/Black individuals with chronic low back pain.
  Interventions: Other: QST
- Caucasian/White QST: This group will consist of a full range of socioeconomic status in Caucasian/White individuals with chronic low back pain.
  Interventions: Other: QST

INTERVENTIONS:
Other: QST — All participants will undergo quantitative sensory testing for assessment of endogenous pain modulation using painful heat, mechanical, and cold stimuli in a laboratory session lasting approximately 1 hour.

SUMMARY:
It remains unclear whether certain disadvantaged subgroups of society may be at heightened risk for poor chronic low back pain (cLBP) outcomes. The overall aim of this study is to incorporate a socioeconomic framework to characterize racial differences in cLBP severity and disability. Further, guided by the theory of fundamental causes, we aim to examine racial and socioeconomic status differences in biopsychosocial predictors of cLBP outcomes, particularly endogenous pain modulation.

DETAILED DESCRIPTION:
Experimental session 1

Resting Blood Pressure and Body Mass Index will be assessed. Participants will complete the Rapid Estimation of Adult Literacy Measure-Short Form (REALM-SF) to determine health literacy. Participants will complete multiple questionnaires to measure Socioeconomic Status, Clinical Pain Assessment and Depression Scale. All participants will undergo quantitative sensory testing for assessment of endogenous pain modulation using painful heat, mechanical, and cold stimuli in a laboratory session lasting approximately 1 hour.

Between Experimental Session 1 and Experimental Session 2

Sleep assessment: Sleep data will be collected by participants in their own homes using objective and subjective measures of their sleep. Participant instructions for how to collect and record their own sleep data will be provided at the end of study session 1.

Experimental Session 2

Experimental session 2 will take place in the CCTS Clinical Research Unit (CRU) All blood will be collected as part of a single draw by research nurses. Participants will complete multiple questionnaires to measure Clinical Pain Assessment and Coping Strategies. Participants will then complete a battery of ecologically valid movement tasks that include: 1) getting in and out of a bed; 2) sitting in a chair, transitioning to a standing position, and then sitting again, and 3) lifting, Performance Battery (SPPB) and the Timed Up and Go test (TUG). Blood will be processed and stored and then used to measure Vitamin D, CRP assays and Oxytocin. Finally follow up data will be collected by phone once per week for four weeks following the completion of study session 2.

ELIGIBILITY:
Inclusion Criteria:

* Chronic low back pain that has been going on consistently for the last 6 months.

Exclusion Criteria:

* Surgery (fusion, Laminectomy) in the last year, accident or trauma in the last year, uncontrolled high blood pressure, heart disease, cancer, diabetes HbA1c > 7%, Ankylosing Spondylitis, Infection, Parkinson's Disease, Multiple Sclerosis, Epilepsy, Stroke, Seizure (non-epileptic), Systemic Lupus Erythematosus, Fibromyalgia, Raynaud's disease, Major Depression/Bipolar Disorder, HIV

Ages: 19 Years to 85 Years | Sex: All
Age Groups: Adult, Older Adult
Gender Based: Yes — Biological gender of either male or female.
Study Population: Men and woman white Caucasian and African American with Chrionic low back pain between the ages of 19-85.
Sampling Method: Non-Probability Sample
Enrollment: 281 (Actual)
Dates: Start 2017-10-15 (Actual); Primary Completion 2024-01-31 (Actual); Study Completion 2024-01-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Burel Goodin, PhD, Principal Investigator — University of Alabama at Birmingham Department of Psychology
Locations (1):
- UAB, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Thomas PA, Ditta PV, Stocking SQ, Webb C, Meints SM, Owens MA, Quinn T, Aroke EN, Morris MC, Sorge RE, Goodin BR, Overstreet DS. The effects of neighborhood disadvantage and adverse childhood experiences on conditioned pain modulation in adults with chronic low back pain. J Pain. 2025 Dec;37S:105566. doi: 10.1016/j.jpain.2025.105566. Epub 2025 Dec 9. PMID 41381165
- [Derived] Thomas PA, Ditta PV, Stocking SQ, Webb C, Meints SM, Owens MA, Quinn T, Aroke EN, Morris MC, Sorge RE, Goodin BR, Overstreet DS. The effects of neighborhood disadvantage and adverse childhood experiences on conditioned pain modulation in adults with chronic low back pain. J Pain. 2025 Jan;26:104706. doi: 10.1016/j.jpain.2024.104706. Epub 2024 Oct 16. PMID 39424112
- [Derived] Thomas PA, Goodin BR, Meints SM, Owens MA, Wiggins AM, Quinn T, Long L, Aroke EN, Morris MC, Sorge RE, Overstreet DS. Adverse Childhood Experiences and Chronic Low Back Pain in Adulthood: The Role of Emotion Regulation. J Pain. 2024 Sep;25(9):104551. doi: 10.1016/j.jpain.2024.104551. Epub 2024 Apr 29. PMID 38692399
- [Derived] Overstreet DS, Strath LJ, Sorge RE, Thomas PA, He J, Wiggins AM, Hobson J, Long DL, Meints SM, Aroke EN, Goodin BR. Race-specific associations: inflammatory mediators and chronic low back pain. Pain. 2024 Jul 1;165(7):1513-1522. doi: 10.1097/j.pain.0000000000003154. Epub 2024 Feb 6. PMID 38323608

RESULTS

PARTICIPANT FLOW:
Period: Year One to Year Two
Arm/Group | African American/Black QST | Caucasian/White QST
Started | 173 | 108
Completed | 165 | 107
Not Completed | 8 | 1
Not completed — High Blood Pressure | 7 | 1
Not completed — HIV + | 1 | 0
Period: Year Two to Year Four
Arm/Group | African American/Black QST | Caucasian/White QST
Started | 165 | 107
Completed | 162 | 107
Not Completed | 3 | 0
Not completed — High Blood Pressure | 1 | 0
Not completed — HIV + | 2 | 0
Period: Year Four to Year Six
Arm/Group | African American/Black QST | Caucasian/White QST
Started | 162 | 107
Completed | 160 | 106
Not Completed | 2 | 1
Not completed — High Blood Pressure | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | African American/Black QST | Caucasian/White QST | Total
Number analyzed (Participants) | 173 | 108 | 281
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 165 | 99 | 264
  >=65 years | 8 | 9 | 17
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 98 | 62 | 160
  Male | 75 | 46 | 121
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 173 | 0 | 173
  White | 0 | 108 | 108
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 173 | 108 | 281
Brief Pain Inventory-Short Form (BPI) pain severity scale [Mean (Standard Deviation); unit: units on a scale] — The BPI pain severity outcome is comprised of four items that assess participants' average, least, and worst pain over the past 24hours, as well as current pain (0=no pain, 10=pain as bad as you can imagine). These 4 items were averaged for a total score (range: 0-10).
  units on a scale | 5.1 (2.1) | 3.9 (1.7) | 4.7 (2.1)

OUTCOME MEASURES:

1. Primary Outcome: Average Clinical Pain Severity
Description: The Brief Pain Inventory Short-Form (BPI-SF) was used to assess clinical pain severity. Four items assessed participants' average, least, and worst pain over the past 24hours, as well as current pain (0=no pain, 10=pain as bad as you can imagine). These 4 items were averaged for a total score (range: 0-10).
Time Frame: Baseline to one week.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | African American/Black QST | Caucasian/White QST
Number analyzed (Participants) | 154 | 96
units on a scale | 5.1 (2.1) | 3.9 (1.7)

2. Secondary Outcome: Average Pain Threshold (Heat)
Description: Pain threshold refers to the intensity at which a stimulus is first perceived as painful. Heat stimuli will be delivered using a computer-controlled thermal stimulation system with a 30 millimeter X 30 millimeter probe. From a baseline of 32 degrees Celsius, the probe temperature will increase at a rate of .5 degrees Celsius/second until the participant responds by pressing a button on a handheld device. For heat pain threshold, participants will be instructed to press the button when the sensation "first becomes painful". Heat pain threshold was assessed at the lumbar spine. On a scale of 32 degrees Celsius to 51 degrees Celsius, with 51 being the hottest temperature.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: degrees Celsius
Arm/Group | African American/Black QST | Caucasian/White QST
Number analyzed (Participants) | 159 | 99
degrees Celsius | 39.96 (13.87) | 40.54 (14.45)

3. Secondary Outcome: Average Pain Tolerance (Heat)
Description: Pain tolerance refers to the maximum amount of pain produced by a stimulus that a person is able/willing to tolerate. Heat stimuli will again be delivered using the computer-controlled thermal stimulation system. From a baseline of 32 degrees Celsius, the probe temperature will increase at a rate of .5 degrees Celsius/second until the participant responds by pressing a button on a handheld device. For heat pain tolerance, participants will be instructed to press the button when they are "no longer willing to tolerate" the painful sensation. Heat pain tolerance was assessed at the lumbar spine. Scale range from 32 degrees Celsius to 51 degrees Celsius with 51 being the hottest.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: degrees Celsius
Arm/Group | African American/Black QST | Caucasian/White QST
Number analyzed (Participants) | 159 | 99
degrees Celsius | 42.50 (13.79) | 44.61 (14.80)

4. Secondary Outcome: Difference in Temporal Summation of Pain (Mechanical)
Description: Temporal summation of pain refers to a form of endogenous pain facilitation characterized by the perception of increased pain despite constant or even reduced peripheral afferent input. Temporal summation is presumed to be the psychophysical manifestation of wind-up. Wind-up is a phenomenon where repetitive stimulation of C primary afferents at rates greater than 0.3 Hertz produces a slowly increasing response of second-order neurons in the spinal cord. Temporal summation was assessed at the lumbar spine using a 512 milliNewton punctate probe. Participants are stimulated once with the punctate probe and asked to provide a pain rating from 0-100 whereby 0 = no pain and 100 = most intense pain imaginable. They are then stimulated 10 consecutive times with the punctate probe and asked to provide another pain rating from 0-100. Temporal summation is the difference between these two ratings, such that positive scores indicate pain facilitation and negative scores indicate pain inhibition.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | African American/Black QST | Caucasian/White QST
Number analyzed (Participants) | 157 | 98
units on a scale | 20.16 (27.64) | 12.68 (18.08)

5. Secondary Outcome: Difference in Pressure Pain Thresholds Assessed Using Conditioned Pain Modulation
Description: Pressure was manually applied and increased at a rate of 30 kPa/s. Participants indicated when the pressure was first perceived to be painful (pressure pain threshold) via button-push. Three applications of a handheld algometer were used to determine baseline pressure pain thresholds (PPTs). Following this, participants underwent two trials of cold pressor immersion. Participants placed their entire hand, up to the wrist, into 12 °C water for 60 s. Immediately following withdrawal of the hand from the cold pressor, the algometer was re-applied at the lumbar region. Participants again indicated when they first perceived the pressure as painful (conditioned PPT). The trial was repeated following a two-minute rest period. The baseline PPTs were averaged, as were the two conditioned PPTs. Conditioned pain modulation was calculated as the difference between Conditioned PPT - Baseline PPT. Positive difference scores indicate pain inhibition and negative scores indicate facilitation.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: Difference in kiloPascals of pressure
Arm/Group | African American/Black QST | Caucasian/White QST
Number analyzed (Participants) | 160 | 97
Difference in kiloPascals of pressure | -7.82 (30.05) | -10.80 (27.43)

6. Secondary Outcome: Total Level of C-reactive Protein
Description: A single blood draw was collected from each participant during their one week follow up visit. The blood was processed and serum was used to quantify C-reactive protein, which is a marker of systemic pro-inflammation. Increasing levels of C-reactive protein are suggestive of greater inflammation.
Time Frame: One week follow up
Measure: Mean (Standard Deviation); unit: nanograms per milliliter
Arm/Group | African American/Black QST | Caucasian/White QST
Number analyzed (Participants) | 155 | 95
nanograms per milliliter | 6394.52 (12828.45) | 5040.71 (5309.51)

7. Secondary Outcome: Total Level of Fibrinogen
Description: Fibrinogen is a protein that plays a crucial role in blood clotting. It is produced by the liver and is present in the blood plasma. Fibrinogen is considered a key player in inflammation, acting as a pro-inflammatory molecule by directly interacting with immune cells and promoting their migration to the site of injury, essentially serving as a "scaffold" for the inflammatory response, and its levels significantly increase during inflammatory conditions, making it a marker for inflammation in the body; high fibrinogen levels often indicate an ongoing inflammatory process.
Time Frame: One week follow up
Measure: Mean (Standard Deviation); unit: nanograms per milliliter
Arm/Group | African American/Black QST | Caucasian/White QST
Number analyzed (Participants) | 131 | 81
nanograms per milliliter | 1656.55 (1052.78) | 1417.26 (1046.08)

8. Secondary Outcome: Total Level of Serum Amyloid A
Description: Serum amyloid A (SAA) is considered a key marker of inflammation, as its levels significantly increase in the blood during an inflammatory response, acting as an "acute phase reactant" produced by the liver when stimulated by pro-inflammatory cytokines like interleukin-6 (IL-6); essentially, high SAA levels indicate the presence of active inflammation in the body.
Time Frame: One week follow up
Measure: Mean (Standard Deviation); unit: nanograms per milliliter
Arm/Group | African American/Black QST | Caucasian/White QST
Number analyzed (Participants) | 131 | 81
nanograms per milliliter | 12224.88 (17436.72) | 9109.35 (12349.25)

9. Secondary Outcome: Total Level of Vitamin D
Description: Vitamin D (also referred to as calciferol) is a fat-soluble vitamin that is naturally present in a few foods, added to others, and available as a dietary supplement. It is also produced endogenously when ultraviolet (UV) rays from sunlight strike the skin and trigger vitamin D synthesis. We quantified Vitamin D from blood serum. Lower levels of Vitamin D have been associated with greater musculoskeletal pain severity and worse bone and muscle health.
Time Frame: One week follow up
Measure: Mean (Standard Deviation); unit: nanograms per milliliter
Arm/Group | African American/Black QST | Caucasian/White QST
Number analyzed (Participants) | 97 | 59
nanograms per milliliter | 20.5 (11.1) | 26.9 (10.3)

10. Secondary Outcome: Total Level of Oxytocin
Description: Oxytocin is a hormone that plays a crucial role in various physiological and behavioral processes, particularly in reproduction, social bonding, and emotional well-being.
Time Frame: One week follow up
Measure: Mean (Standard Deviation); unit: nanograms per milliliter
Arm/Group | African American/Black QST | Caucasian/White QST
Number analyzed (Participants) | 51 | 38
nanograms per milliliter | 181.54 (69.39) | 192.71 (87.92)

11. Secondary Outcome: Sleep Quality
Description: Insomnia Severity Index (ISI) was used to measure sleep quality. The ISI is a seven-item questionnaire used to evaluate the severity and impact of insomnia. Participants used a 5-point Likert scale to rate severity of difficulties with sleep onset and sleep maintenance as well as problems with early morning awakenings, sleep dissatisfaction, and interference of sleep difficulties with daytime functioning within the last month. Items are summed to calculate a total score ranging from 0 to 28, thus, indicating absence of insomnia (0-7), subthreshold insomnia (8-14), moderate insomnia (15-21) and severe insomnia (22-28).
Time Frame: Between baseline and one week follow-up
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | African American/Black QST | Caucasian/White QST
Number analyzed (Participants) | 155 | 97
units on a scale | 12.08 (7.10) | 12.12 (7.40)

12. Secondary Outcome: Self-reported Disability
Description: Self-reported disability was assessed using the Graded Chronic Pain Scale (GCPS) - interference scale. A higher score on the interference section indicates a greater level of disruption to daily life due to pain. The GCPS scale ranges from 0-100 and higher scores are indicative of greater self-reported disability.
Time Frame: One week follow up
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | African American/Black QST | Caucasian/White QST
Number analyzed (Participants) | 155 | 96
units on a scale | 53.40 (29.49) | 41.96 (26.39)

13. Secondary Outcome: Evoked Pain With Movement
Description: The Short Physical Performance Battery was used to assess movement-evoked pain. Participants completed three movements (balance, chair stands, and walking). After completion of each movement task, participants were asked to provide a pain intensity rating for any movement-evoked pain experienced during completion of the balance, chair stands, and walking tests. The 0-100 numeric rating scale was utilized for this purpose, whereby: (0 = no pain and 100 = most intense pain imaginable). Average pain intensity was calculated across the three movements.
Time Frame: One week follow up
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | African American/Black QST | Caucasian/White QST
Number analyzed (Participants) | 159 | 99
units on a scale | 31.01 (31.00) | 13.33 (18.88)

14. Secondary Outcome: Functional Performance
Description: The Short Physical Performance Battery (SPPB) is an objective measurement instrument of balance, lower extremity strength, and functional capacity in adults. The test includes three different domains (walking, sit-to-stand and balance) to assess functional mobility. Scores range from 0 to 12 with higher scores suggest of better functional performance.
Time Frame: One week follow up
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | African American/Black QST | Caucasian/White QST
Number analyzed (Participants) | 159 | 99
units on a scale | 8.95 (1.81) | 9.82 (1.75)

15. Other Pre Specified Outcome: Depressive Symptoms
Description: The 20-item Center for Epidemiological Studies- Depression (CES-D) scale was used to measure depressive symptoms over the past week (0=rarely or none of the time [less than 1 day], 3=most or all of the time [5-7days]). All items were summed, such that higher scores suggest greater depression severity (range: 0-60).
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | African American/Black QST | Caucasian/White QST
Number analyzed (Participants) | 154 | 96
units on a scale | 16.0 (10.0) | 17.6 (11.8)

16. Other Pre Specified Outcome: Average Perceived Injustice (Pain-related)
Description: The Injustice Experience Questionnaire (IEQ) was used to assess perception of pain-related injustice in this sample. Participants rated the frequency with which they experienced each of 12 thoughts/feelings when reflecting on their chronic pain condition. Items are rated on a scale of 0 (never) to 4 (all of the time). Injustice Experience Questionnaire items broadly reflect the associated factors of "severity/irreparability of loss" and "blame/unfairness." Representative severity/irreparability items include "Most people don't understand how severe my condition is, and "My life will never be the same." Blame/unfairness items include "I am suffering because of someone else's negligence, and "It all seems so unfair." The total score was used and it ranges from 0 to 48 with higher scores representing greater perceived injustice.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | African American/Black QST | Caucasian/White QST
Number analyzed (Participants) | 159 | 95
units on a scale | 15.69 (12.68) | 13.85 (11.50)

17. Other Pre Specified Outcome: Perceived Discrimination
Description: The Experiences of Discrimination (EOD) scale was used to assess lifetime occurrences of racial discrimination across 9 different domains (eg, at work, getting medical care). Participants rated the frequency with which they perceived experiencing discrimination in each situation (0=never, 1=once, 2.5=2-3 times, 5=4 or more times). Responses across all items were summed and higher score suggest greater perceived discrimination (range: 0-45).
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | African American/Black QST | Caucasian/White QST
Number analyzed (Participants) | 154 | 96
units on a scale | 10.3 (9.6) | 4.1 (8.1)

18. Other Pre Specified Outcome: Social Support
Description: Measured using the Multidimensional Survey of Perceived Social Support Scale (MSPSS). This scale consisted of 12 items that measure the extent of social support received from 3 specific sources: friends, family, and significant others. Types of social support assessed by the MSPSS included emotional (eg, "I get the emotional help and support I need from my family"), tangible (eg, "There is a special person who is around when I am in need"), informational (eg, "My family is willing to help me make decisions"), social network support (eg, "I can count on my friends when things go wrong"), and esteem (eg, "I have a special person who is a real source of comfort to me"). Each item was scored on a scale ranging from 1 (very strongly disagree) to 7 (very strongly agree). Summation of the 12 item scores provided a possible total score ranging from 12 to 84 for overall social support, with higher scores corresponding to higher levels of social support.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | African American/Black QST | Caucasian/White QST
Number analyzed (Participants) | 154 | 95
units on a scale | 64.62 (15.60) | 65.88 (15.01)

19. Other Pre Specified Outcome: Total Psychological Pain Resilience
Description: The Pain Resilience Scale (PRS) is a 14-item assessment of resilience in the presence of intense or prolonged pain. The assessment has 2 subscales to measure specific domains of resilience: behavioral perseverance and cognitive/affective positivity. The behavioral perseverance subscale examines an individual's ability to continue engaging in behaviors or activity when experiencing pain. The cognitive/affective positivity subscale examines an individual's ability to maintain positive thoughts and manage negative thoughts or emotions while in pain. Each item is scored from 0 (not at all) to 4 (all the time) to determine the degree to which individuals engage in resiliency resources. The total Pain Resilience Scale (PRS) ranges from 0 to 56, calculated as the sum of all 14 items. Higher scores suggest greater pain resilience.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | African American/Black QST | Caucasian/White QST
Number analyzed (Participants) | 159 | 96
units on a scale | 39.49 (10.41) | 38.82 (10.13)

20. Other Pre Specified Outcome: Average Dietary Caffeine Consumption
Description: Measured using a daily diary of dietary intake across seven days. The value presented represents the average daily caffeine consumption.
Time Frame: Between baseline and one week follow up
Measure: Mean (Standard Deviation); unit: milligrams per day
Arm/Group | African American/Black QST | Caucasian/White QST
Number analyzed (Participants) | 31 | 31
milligrams per day | 165.12 (208.10) | 219.13 (208.49)

ADVERSE EVENTS:
Time Frame: 6 weeks
Description: We had no adverse events linked to this protocol.
Arm/Group | African American/Black QST | Caucasian/White QST
All-Cause Mortality (participants affected / at risk) | 0/173 | 0/108
Serious Adverse Events (participants affected / at risk) | 0/173 | 0/108
Other Adverse Events (participants affected / at risk) | 15/173 | 1/108
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | African American/Black QST (N=173) | Caucasian/White QST (N=108)
High Blood Pressure (Cardiac disorders) | 12 (12) | 1 (1)
HIV + (Immune system disorders) | 3 (3) | 0 (0)

LIMITATIONS AND CAVEATS:
Due to a delay in the initial award notification, start up was delayed in the first year. Recruitment increased and the protocol infrastructure was complete when the Covid 19 pandemic stopped all protocol recruitment and all study tasks. After the pandemic, recruitment was slower, the study timeline indicated recruitment completion at the end of 2022, but we had to request a No Cost Extension from January 2022 to January 2023 to complete recruitment numbers.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-12-18): https://cdn.clinicaltrials.gov/large-docs/92/NCT03338192/Prot_SAP_000.pdf